CLINICAL TRIAL: NCT04279600
Title: Taurine Supplementation and Physical Training Effects on Adipose Tissue Mitochondrial Energy Metabolism, and Blood Inflammation and Oxidative Stress in Obese Women
Brief Title: Taurine Supplementation and Training Effects on Energy Metabolism, Inflammation and Oxidative Stress in Obese Women
Acronym: Taurine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Taurine
Record Dates: First submitted 2019-08-18; First posted 2020-02-21 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Taurine; Exercise

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Supplement capsule packages were labeled as "Supplement A" and "Supplement B" and the nutrient (taurine or placebo- starch) was revealed after the end of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Taurine supplementation (Experimental): Taurine supplementation composed of capsules of taurine powder. Dosage: 3 grams/day Frequency: 1 time/day Duration: 8 weeks
  Interventions: Dietary Supplement: Taurine
- Taurine supplementation associated to exercise training (Active Comparator): Taurine supplementation composed of capsules of taurine powder. Dosage: 3 grams/day Frequency: 1 time/day Duration: 8 weeks
  Exercise training Exercise Protocol: a combination of strength and aerobic exercises Duration: 2 weeks of adaptation and 8 weeks of physical training. Frequency: 3 times/week Duration: 55 minutes/session Intensity: 75 to 90% of maximum heart rate
  Interventions: Dietary Supplement: Taurine; Other: Exercise training
- Placebo supplementation associated to exercise training (Placebo Comparator): Placebo supplementation composed of capsules of starch powder. Dosage: 3 grams/day Frequency: 1 time/day Duration: 8 weeks
  Exercise training Exercise Protocol: a combination of strength and aerobic exercises Duration: 2 weeks of adaptation and 8 weeks of physical training. Frequency: 3 times/week Duration: 55 minutes/session Intensity: 75 to 90% of maximum heart rate
  Interventions: Dietary Supplement: Placebo; Other: Exercise training

INTERVENTIONS:
Dietary Supplement: Taurine — Taurine supplementation in capsules of 1 gram of taurine powder, total dosage: 3 grams/day
  Arms: Taurine supplementation; Taurine supplementation associated to exercise training
Dietary Supplement: Placebo — Placebo supplementation in capsules of 1 gram of starch powder, total dosage: 3 grams/day
  Arms: Placebo supplementation associated to exercise training
Other: Exercise training — 4 weeks of combined exercise training (alternating strength and aerobic exercise), with a frequency of 3 times/week with 55 min/day.
  Arms: Placebo supplementation associated to exercise training; Taurine supplementation associated to exercise training

SUMMARY:
Taurine supplementation researches have increased due to its antioxidant and anti-inflammatory actions, and its ability to modulate lipid metabolism by stimulating the expression of proteins that regulates mitochondrial biogenesis and increases respiratory function (PGC-1α and PPAR) and irisin release when associated to exercise. Since obesity can induce metabolic disorders including abnormal production of adipokines and activation of pro-inflammatory signaling pathways also mitochondrial metabolism dysfunction in the adipose tissue, the use of taurine would be a new strategy for obesity prevention and treatment. Moreover, the association of taurine and exercise could improve exercise effects, promote higher energy expenditure and increase mitochondrial respiration, consequently resulting in weight loss. Therefore, the present investigation aims to evaluate the effects of the association of taurine supplementation and a combined exercise training protocol (aerobic and strength) on resting energy expenditure, weight, body composition, blood markers of inflammation and oxidative stress, telomeres length, and mitochondrial function and the expression of genes that regulates energy metabolism and lipid oxidation in the white adipose tissue in obese women.

DETAILED DESCRIPTION:
A double-blind placebo-controlled study was conducted with 24 obese women (32.9±6.3 years). Capsules of taurine (3 grams) (GTau) or placebo (GP) were daily supplemented 2 hours before training. The training program was composed of aerobic and strength exercises during one hour, 3 times a week, for an 8-week period (intensity of 80% heart rate). The taurine supplemented group received only taurine capsules (3g/day) during 8 weeks. Measurement of weight, hip and waist circumference, and body composition (by Deuterium oxide) were performed before and after the intervention. Resting energy expenditure and nutrients oxidation were assessed by calorimetry.

In order to check the effects of the intervention, abdominal tissue biopsy will be performed for white adipose tissue analysis, evaluation of mitochondrial function and quantification of the expression of genes related to energy metabolism and lipid oxidation and taurine pathway; blood collection will be done for quantification of taurine levels, inflammatory (IL-10, IL-15, IL-6, IL-1, TNF-α, and CRP), adipokines (adiponectin, adipsin, resistin, fetuin and leptin) and oxidative stress (GPx, SOD and MDA) markers. Also, evaluation of telomere length was performed. Body composition was evaluated by deuterium oxide method, weight, waist and hip circumference were accessed. All the measurements were performed before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 30 to 40 kg / m²
* Sedentary
* No associated co morbidity

Exclusion Criteria:

* Women who have a medical impediment to the practice of physical exercise
* Women that have undergone bariatric surgery
* Menopause, cancer or any metabolic disease
* Smokers
* Alcoholics
* Insulin-dependent diabetes

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in white adipose tissue mitochondrial respiration at 8 weeks | eight weeks
  A subcutaneous adipose tissue sample collected for analysis of mitochondrial respiration (mitochondrial uncoupled state, phosphorylation state and electron transport system maximal capacity) were calculated at 8 weeks in comparison to the baseline.
Change from baseline in indirect calorimetry at 8 weeks | eight weeks
  Change of energy expenditure and lipids oxidation were calculated at 8 weeks in comparision to the baseline.
Changes from baseline in interleukines levels at 8 weeks | eight weeks
  Change of inflammatory markers such as interleukines 6, 10 and 15 were calculated at 8 weeks in comparision to the baseline.
Changes from baseline in cytokine levels at 8 weeks | eight weeks
  Change of inflammatory markers such as adiponectin, resistin and adipsin were calculated at 8 weeks in comparision to the baseline.
Changes from baseline in glutathione peroxidase levels at 8 weeks | eight weeks
  Change of oxidative stress markers such as glutathione peroxidase were calculated at 8 weeks in comparision to the baseline.
Changes from baseline in superoxide dismutase levels at 8 weeks | eight weeks
  Change of oxidative stress markers such as superoxide dismutase were calculated at 8 weeks in comparision to the baseline.
Changes from baseline in macronutrient intake at 8 weeks | eight weeks
  Change of macronutrient intake were calculated at 8 weeks in comparision to the baseline.
Changes from baseline in total calorie intake at 8 weeks | eight weeks
  Change of total calorie intake were calculated at 8 weeks in comparision to the baseline.
Changes from baseline in body composition at 8 weeks | eight weeks
  Change of body composition through deuterium oxide method were calculated at 8 weeks in comparision to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen C Freitas, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Physical Education and Sport of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bostrom P, Wu J, Jedrychowski MP, Korde A, Ye L, Lo JC, Rasbach KA, Bostrom EA, Choi JH, Long JZ, Kajimura S, Zingaretti MC, Vind BF, Tu H, Cinti S, Hojlund K, Gygi SP, Spiegelman BM. A PGC1-alpha-dependent myokine that drives brown-fat-like development of white fat and thermogenesis. Nature. 2012 Jan 11;481(7382):463-8. doi: 10.1038/nature10777. PMID 22237023
- [Background] Ghandforoush-Sattari M, Mashayekhi S, Krishna CV, Thompson JP, Routledge PA. Pharmacokinetics of oral taurine in healthy volunteers. J Amino Acids. 2010;2010:346237. doi: 10.4061/2010/346237. Epub 2010 Jun 29. PMID 22331997
- [Background] Heilbronn LK, Gan SK, Turner N, Campbell LV, Chisholm DJ. Markers of mitochondrial biogenesis and metabolism are lower in overweight and obese insulin-resistant subjects. J Clin Endocrinol Metab. 2007 Apr;92(4):1467-73. doi: 10.1210/jc.2006-2210. Epub 2007 Jan 23. PMID 17244782
- [Background] Kraunsoe R, Boushel R, Hansen CN, Schjerling P, Qvortrup K, Stockel M, Mikines KJ, Dela F. Mitochondrial respiration in subcutaneous and visceral adipose tissue from patients with morbid obesity. J Physiol. 2010 Jun 15;588(Pt 12):2023-32. doi: 10.1113/jphysiol.2009.184754. Epub 2010 Apr 26. PMID 20421291
- [Background] Lourenco R, Camilo ME. Taurine: a conditionally essential amino acid in humans? An overview in health and disease. Nutr Hosp. 2002 Nov-Dec;17(6):262-70. PMID 12514918
- [Background] Marion-Latard F, Crampes F, Zakaroff-Girard A, De Glisezinski I, Harant I, Stich V, Thalamas C, Riviere D, Lafontan M, Berlan M. Post-exercise increase of lipid oxidation after a moderate exercise bout in untrained healthy obese men. Horm Metab Res. 2003 Feb;35(2):97-103. doi: 10.1055/s-2003-39051. PMID 12734789
- [Background] de Almeida Martiniano AC, De Carvalho FG, Marchini JS, Garcia SB, Junior JE, Mauad FM, da Silva AS, de Moraes C, de Freitas EC. Effects of taurine supplementation on adipose tissue of obese trained rats. Adv Exp Med Biol. 2015;803:707-14. doi: 10.1007/978-3-319-15126-7_56. No abstract available. PMID 25833538
- [Background] Schuller-Levis GB, Park E. Taurine: new implications for an old amino acid. FEMS Microbiol Lett. 2003 Sep 26;226(2):195-202. doi: 10.1016/S0378-1097(03)00611-6. PMID 14553911
- [Background] Suzuki T, Suzuki T, Wada T, Saigo K, Watanabe K. Taurine as a constituent of mitochondrial tRNAs: new insights into the functions of taurine and human mitochondrial diseases. EMBO J. 2002 Dec 2;21(23):6581-9. doi: 10.1093/emboj/cdf656. PMID 12456664
- [Background] Tsuboyama-Kasaoka N, Shozawa C, Sano K, Kamei Y, Kasaoka S, Hosokawa Y, Ezaki O. Taurine (2-aminoethanesulfonic acid) deficiency creates a vicious circle promoting obesity. Endocrinology. 2006 Jul;147(7):3276-84. doi: 10.1210/en.2005-1007. Epub 2006 Apr 20. PMID 16627576
- [Background] Yin X, Lanza IR, Swain JM, Sarr MG, Nair KS, Jensen MD. Adipocyte mitochondrial function is reduced in human obesity independent of fat cell size. J Clin Endocrinol Metab. 2014 Feb;99(2):E209-16. doi: 10.1210/jc.2013-3042. Epub 2013 Nov 25. PMID 24276464
- [Background] Zhang M, Izumi I, Kagamimori S, Sokejima S, Yamagami T, Liu Z, Qi B. Role of taurine supplementation to prevent exercise-induced oxidative stress in healthy young men. Amino Acids. 2004 Mar;26(2):203-7. doi: 10.1007/s00726-003-0002-3. Epub 2003 May 9. PMID 15042451
- [Derived] De Carvalho FG, Brandao CFC, Munoz VR, Batitucci G, Tavares MEA, Teixeira GR, Pauli JR, De Moura LP, Ropelle ER, Cintra DE, da Silva ASR, Junqueira-Franco MVM, Marchini JS, De Freitas EC. Taurine supplementation in conjunction with exercise modulated cytokines and improved subcutaneous white adipose tissue plasticity in obese women. Amino Acids. 2021 Sep;53(9):1391-1403. doi: 10.1007/s00726-021-03041-4. Epub 2021 Jul 13. PMID 34255136